CLINICAL TRIAL: NCT05055479
Title: Nosocomial Outbreak of Monoclonal VIM Carbapenemase Producing Enterobacter Cloacae in an Intensive Care Unit During SARS-CoV-2 Pandemic
Brief Title: Nosocomial Outbreak of BHRe in an Intensive Care Unit During SARS-CoV-2 Pandemic
Acronym: BHReICU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0187
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Enterobacteriaceae Infections; Hospital-Acquired Infection
Keywords: outbreak; Enterobacteriaceae Infections; Hospital-Acquired Infection; integrated approach; VIM
MeSH Terms: conditions — Enterobacteriaceae Infections; Cross Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multidrug Resistant (MDR) bacteria have become a major worldwide public health challenge and hospitals are now increasingly faced with management of local outbreaks involving such pathogens. Especially, intensive care units (ICU) provide an ideal background for outbreaks caused by MDR bacteria among which carbapenemase-producing Enterobacteriaceae (CPE) can be found. Among CPE involved in ICU outbreaks, VIM producers have been reported worldwide, and described as especially difficult to control. The COVID-19 pandemic and all of the measures health workers have to implement to fight the spread of SARS-Cov-2 have also impacted the management of such outbreaks. In this retrospective study, the investigators aim to describe the management of an outbreak caused by a VIM-producing Enterobacter cloacae strain during the 2020 COVID-19 pandemic in an ICU, and show the importance of concerted measures and actions implemented at multiple levels to prevent the spread of this MDR strain.

DETAILED DESCRIPTION:
Multidrug Resistant (MDR) bacteria have become a major worldwide public health challenge and hospitals are now increasingly faced with management of local outbreaks involving such pathogens. Especially, intensive care units (ICU) provide an ideal background for outbreaks caused by MDR bacteria among which carbapenemase-producing Enterobacteriaceae (CPE) can be found. Among CPE involved in ICU outbreaks, VIM producers have been reported worldwide, and described as especially difficult to control. The COVID-19 pandemic and all of the measures health workers have to implement to fight the spread of SARS-Cov-2 have also impacted the management of such outbreaks. The likely source of an outbreak is not always easy to pinpoint, but some common sources can be cited: an index patient with a history of hospitalization abroad, a contaminated instrument, and/or an environmental reservoir. CPE outbreaks in ICU usually have multifactorial origins, thus needing to combine several actions to be controlled. Infection and prevention control (IPC) measures habitually rely on patients screening, use of contact precautions, staff education, enhanced environmental cleaning, cohorting of patients and staff as well as a proper antimicrobial stewardship. Investigation of these outbreaks and implementation of IPC measures are ensured by various professional categories in the hospital. This implies a tight cooperation and communication between all involved healthcare workers.

In this retrospective study, the investigators aim to describe the management of an outbreak caused by a VIM-producing Enterobacter cloacae strain during the 2020 COVID-19 pandemic in an ICU, and show the importance of concerted measures and actions implemented at multiple levels to prevent the spread of this MDR strain.

ELIGIBILITY:
Inclusion Criteria:

* patients who have stayed in ICU
* patients with positive sample to E. cloacae VIM between March and October 2020

Exclusion Criteria:

* patients who didn't agreed to be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have stayed in ICU and with positive sample to E. cloacae VIM between March and October 2020.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Change in care type of BHRe in ICU | 1 month
  Management of VIM-producing Enterobacter cloacae strain care in ICU.
  All types of therapeutics used to manage atrial fibrillation are collected

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mullie C, Lemonnier D, Adjide CC, Maizel J, Mismacque G, Cappe A, Carles T, Pierson-Marchandise M, Zerbib Y. Nosocomial outbreak of monoclonal VIM carbapenemase-producing Enterobacter cloacae complex in an intensive care unit during the COVID-19 pandemic: an integrated approach. J Hosp Infect. 2022 Feb;120:48-56. doi: 10.1016/j.jhin.2021.11.017. Epub 2021 Nov 30. PMID 34861315